CLINICAL TRIAL: NCT05438680
Title: Evaluation of the Effect of Bovine Colostrum in Prevention of Late Onset Sepsis and Retinopathy of Prematurity
Brief Title: Bovine Colostrum in Prevention of Sepsis and Retinopathy of Prematurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Farag, Primary Investigator and Lecturer in Pediatrics, Faculty of Medicine, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0106797
Record Dates: First submitted 2022-06-13; First posted 2022-06-30 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Preterm
Keywords: Premature infants; colostrum; ROP
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Masking controlled clinical trial will be used to assess the effect of prophylactic bovine colostrum in preventing retinopathy of prematurity.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I: bovine colostrum group (Active Comparator)
  Interventions: Dietary Supplement: The bovine colostrum ( trade name : baby steps sachets, 300mg )
- group II : control group (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: The bovine colostrum ( trade name : baby steps sachets, 300mg ) — The bovine colostrum sachets will be used in a dose of 3.5ml/kg/ day , starting from the first 3 days after birth, for 14 days.
  Enteral route, either through nasogastric tube or orally.
  Arms: Group I: bovine colostrum group
Dietary Supplement: Placebo — distilled water with no bovine colostrum
  Arms: group II : control group

SUMMARY:
The aim of this study is to evaluate efficacy of bovine colostrum administration as a prophylaxis to decrease the incidence and the occurrence of retinopathy of prematurity in preterm neonates of gestational age less than 32 weeks during their hospital stay.

DETAILED DESCRIPTION:
This study will include a randomized controlled trial carried out on preterm neonates who will fulfill the eligibility criteria delivered at Alexandria University Children's Hospital. Evaluation of the outcome will be done only for those who admitted to the neonatal intensive care unit (NICU) at Alexandria University Children's Hospital.

The study will be carried out in 4 phases:

1. First phase: Enrollment and selection phase.
2. Second phase: Intervention phase ( enteral bovine colostrum administration) .
3. Third phase: Evaluation phase.
4. Fourth phase: collected data analysis and results.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants ≤ 32 weeks gestational age, weight ≤ 1500 gm. Start feeding in the first 72 hours of life

Exclusion Criteria:

* Exclusion criteria

Patients with any of the following will be excluded:

1. Obvious major congenital abnormalities.
2. Infants expected to be >72 hours of age at the time of randomization.
3. Parental consent lacking/refusal

Ages: 1 Hour to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Fundus examination to detect retinopathy of prematurity | 28 days
  ROP screen will be performed by ophthalmologist to detect zone stage extension and severity of the disease

SECONDARY OUTCOMES:
prematurity related complications | 28 days
  * late onset sepsis
  * IVH
  * Necrotizing enterocolitis
  * bronchopulmonary dysplasia
Assessment of weight | 28 days
  -Assessment of weight every other day.
-Assessment of Head circumference | 28 days
  measurement of Head circumference weekly.
-Assessment of length | 28 days
  -Assessment of length on admission and on discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Alaaaldin Thabet, PhD, Study Director — Faculty of medicine, Alexandria University, Egypt; Islam Shereen Hamdy, PhD, Study Director — Faculty of medicine, Alexandria University, Egypt; Eman Shabban Mohamed, MBBCh, Principal Investigator — Faculty of medicine, Alexandria University, Egypt; Marwa Mohamed Farag, PhD, Study Chair — Faculty of medicine, Alexandria University, Egypt
Locations (2):
- Egypt (2):
  - Alexandria university, Elshattbi hospital, Alexandria
  - Marwa Mohamed Farag, Alexandria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farag MM, Thabet MAEH, Ahmed IS, Hanafi NF, Elsawy WS, Mohamed ES. Do preterm infants' retinas like bovine colostrum? A randomized controlled trial. Ital J Pediatr. 2024 Oct 19;50(1):218. doi: 10.1186/s13052-024-01781-z. PMID 39427215